CLINICAL TRIAL: NCT03461068
Title: The Effect of Exogenous Ketone Monoester Supplement on Glycemic Response to an Oral Glucose Tolerance Test
Brief Title: Exogenous Ketones and Glucose Tolerance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H16-01846
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Ketones; Dietary Supplements
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo masked with flavouring and participants consume in opaque containers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone monoester (Experimental): Acute morning dose of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (0.45 ml/kg body weight)
  Interventions: Dietary Supplement: Ketone monoester
- Placebo (Placebo Comparator): Acute morning dose of flavour-matched placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoester — Acute ingestion of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate prior a 2-hour oral glucose tolerance test.
  Arms: Ketone monoester
Dietary Supplement: Placebo — Acute ingestion of a taste-matched placebo prior a 2-hour oral glucose tolerance test.
  Arms: Placebo

SUMMARY:
The ketone body beta-hydroxybutyrate is produced during prolonged fasting or when endogenous carbohydrate stores are depleted and can be used as an alternative fuel source. Exogenous beta-hydroxybutyrate, in the form of a ketone monoester, is proposed to have glucose-lowering potential but this has not been adequately studied. The purpose of this study is to determine whether supplementing with an acute dose of ketone monoester can improve the glycemic response to an oral glucose tolerance test in individuals with impaired fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

* Not taking any medications affecting glucose metabolism.
* Elevated fasting glucose level (5.6-6.9 mmol/L) OR body mass index >28 kg/m2 OR elevated waist circumference (>102 cm for males, >88 cm for females)

Exclusion Criteria:

* Diagnosed with diabetes.
* Diagnosed with heart disease.
* Competitive endurance athlete (self-identified as engaged in specific endurance training in triathlon, cycling, or distance running and competing in races or competition)
* Recent (last 3 months) or current consumption of a low-carbohydrate ketogenic diet
* Current consumption of ketone supplements
* Pregnant or planning to become pregnant during the study (if female)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve | 2-hour
  Area under the curve for glucose during oral glucose tolerance test

SECONDARY OUTCOMES:
Insulin area under the curve | 2-hour
  Insulin area under the curve during oral glucose tolerance test
Free fatty acids area under the curve | 2-hour
  Non-esterified fatty acids area under the curve during oral glucose tolerance test
Caspase-1 activation | 15 minutes
  Caspase-1 activation assessed before and after ketone or placebo ingestion in the morning
Inflammatory cytokines | 15 minutes
  Inflammatory cytokines assessed before and after ketone or placebo ingestion in the morning
C-peptide area under the curve | 2-hour
  C-peptide area under the curve during oral glucose tolerance test
GLP-1 area under the curve | 2-hour
  GLP-1 area under the curve during oral glucose tolerance test
Glucagon area under the curve | 2-hour
  Glucagon area under the curve during oral glucose tolerance test
Glucose incremental area under the curve | 2-hour
  Incremental area under the curve (above baseline) for glucose during oral glucose tolerance test
Insulin incremental area under the curve | 2-hour
  Incremental area under the curve (above baseline) for insulin during oral glucose tolerance test
2-hr glucose level | 2-hour
  Plasma glucose assessed 2-hr after oral glucose tolerance test.
Oral glucose sensitivity index | 2-hour
  Oral glucose sensitivity index derived from glucose and insulin values throughout the 2-hr oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myette-Cote E, Caldwell HG, Ainslie PN, Clarke K, Little JP. A ketone monoester drink reduces the glycemic response to an oral glucose challenge in individuals with obesity: a randomized trial. Am J Clin Nutr. 2019 Dec 1;110(6):1491-1501. doi: 10.1093/ajcn/nqz232. PMID 31599919